CLINICAL TRIAL: NCT02875418
Title: A Study Aimed at Comparing Two Methods of Contractions Monitoring (Electrical Uterine Monitor - EUM vs. Tocodynamometer) for Clinical Decision Making Regarding Treatment Among Pregnant Women With Preterm Contractions.
Brief Title: Comparing Two Methods of Contractions Monitoring for Clinical Decision Making Regarding Treatment Among Pregnant Women With Preterm Contractions.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 171-16-TLV
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Fetal Heartbeat Tracings
MeSH Terms: interventions — Uterine Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUM and tocodynamometry (Experimental): Pregnant women with gestational age 24+0/7 to 33+6/7 weeks of gestation and contractions, cramping, pelvic pressure or backache.
  Interventions: Device: EUM; Device: Tocodynamometry

INTERVENTIONS:
Device: EUM — STUDY DESIGN
  1. Explanation regarding the study and assessing eligibility criteria.
  2. Signing an informed consent.
  3. Recording of uterine contractions by both EUM and tocodynamometry. A correlation between EUM and tocodynamometry will be calculated. For the purpose of this study, a positive EUM or tocodynamometry will be defined as 3 at least 3 contractions in 30 minutes.
Device: Tocodynamometry — STUDY DESIGN
  1. Explanation regarding the study and assessing eligibility criteria.
  2. Signing an informed consent.
  3. Recording of uterine contractions by both EUM and tocodynamometry. A correlation between EUM and tocodynamometry will be calculated. For the purpose of this study, a positive EUM or tocodynamometry will be defined as 3 at least 3 contractions in 30 minutes.

SUMMARY:
Background:

Identification and measurement of uterine contractions throughout pregnancy and labor is crucial to the well being of both mother and fetus. Prematurity is one of the major causes for adverse pregnancy outcomes, and clinical decision-making often relies on uterine frequency as recorded by a tocodynamometer, as well as on other methods including sonographic cervical length, pelvic examination.

Objective:

To show that the use of the EUM in preterm labor is effective in establishing true preterm labor.

DETAILED DESCRIPTION:
Methods:

Currently, three methods of assessing uterine activity exist. The first, tocodynamometry, is based on mechanical measurement of abdominal wall stiffness by a strain gauge placed externally on the patient's abdomen. This method mainly displays the presence of a contraction, its duration and the frequency of contractions. Yet, it fails to reflect the actual quantity of baseline tone or contraction amplitude due to great variability in placement and the gravida's body habitus. It is also unable to distinguish between true contractions or maternal movements or maternal Valsalva maneuver such as in coughing, straining or sneezing. These are the main reasons this technology is known to be unreliable in many cases and shows high percentage of false positive and false negative results [1].

Another method for monitoring uterine contractions is an internal measurement of uterine pressure via an Intra-Uterine Pressure Catheter (IUPC). While it is accurate in recording intensity, duration and frequency of contractions, as well as uterine basal tone, it has two principle limitations: the IUPC can only be used after rupture of the membranes, and the introduction of a foreign object in the uterine cavity may result in chorioamnionitis.

The third method of evaluating uterine activity involves recording of the myometrial electrical activity [2]. Initially, this was assessed in animal models by means of invasive uterine EMG [3-6], followed by noninvasive EMG recordings from abdominal surface in humans [7-10]. Several studies have attempted to correlate between term and preterm labor to uterine EMG, with limited success [11-17]. However, although most traditional EMG devices use only 2 electrodes, a multichannel, noninvasive EMG device have been used successfully in previous studies, both in preterm and term pregnancies, and were proved as both safe and accurate [18-25]. Recently, reliability studies were published, regarding the comparison to tocodynamomtery, IUPC and electrical uterine monitoring, using a multichannel EMG, and demonstrated the multichannel EMG is as good as the IUPC ('Gold Standard') and both multichannel EMG and IUPC are superior to tocodynamometry in recording uterine activity [26-27].

Study rational Premature labor and delivery heralds great costs to the healthcare system, including admission costs, tocolytic treatment and side effects and neonatal treatment of the preterm neonate. Unfortunately, the accuracy of diagnosing preterm labor is poor, with less than 10% of women presenting with preterm labor symptoms actually delivering within 7 days of symptoms' onset [28], 30% with resolving symptoms and more than 50% delivering at term [29]. Since IUPC cannot be used in women with intact membranes and tocodynamometry is unreliable, with previous reports concluding that multichannel EMG is superior to tocodynamomtery and comparable to IUPC, our objective is to evaluate the utility of the multichannel EMG in women with preterm contractions.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age 24+0/7 to 33+6/7 weeks of gestation.
2. Maternal age > 18 years.
3. Contractions, cramping, pelvic pressure or backache.
4. Reactive fetal heart rate monitoring at enrollment.
5. Subjects are willing and able to comply with the requirements of the protocol.
6. Fully understand all elements of the study, and have signed and dated, the written informed consent form before initiation of protocol-specified procedures.

Exclusion Criteria:

1. Refusal to participate.
2. Maternal age < 18 years.
3. Woman with implanted electronic device of any kind.
4. Woman with allergy to silver.
5. Irritated skin or open wound.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Rate of preterm deliveries | 4 month
  Week of gestation will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: yariv yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No